CLINICAL TRIAL: NCT00466804
Title: Observational Study of Alloimmunity in Cardiac Transplant Recipients
Brief Title: Noninvasive Methods to Monitor Graft Survival in Heart Transplant Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-05
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Heart Transplant
Keywords: heart transplant recipients; organ transplantation; immune biomarkers; transplant rejection
MeSH Terms: interventions — Heart Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples may be retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart Transplant Recipients: People who will have a heart transplant
  Interventions: Procedure: Heart transplant

INTERVENTIONS:
Procedure: Heart transplant — People in this study will have a heart transplant and be monitored for signs of rejection

SUMMARY:
Injury of transplant tissue by a transplant recipient's immune system continues to be the leading cause of graft rejection and recipient death. The purpose of this study is to identify a single test or a combination of noninvasive tests currently used for heart transplant monitoring that correlate to long-term graft survival.

DETAILED DESCRIPTION:
A major cause of heart transplant failure is the blockage of blood flow from lesions caused by ongoing injury and repair of the graft by the host's immune system. However, the role of T cells, antibodies, and other parts of the recipient's immune system are not well understood in transplant injury. Currently, there are no effective, noninvasive ways to detect or predict how an individual's immune system will react to a transplant. The purpose of this study is to correlate current noninvasive monitoring tests with long-term graft survival and function, and determine which tests are the most accurate predictors of this survival.

Participants in this study must currently be on the waiting list for a heart transplant and have a donor heart available to them. This study will consist of six study visits over 12 months. The baseline visit will occur on the day of transplantation. Follow-up visits will occur at Week 6 and Months 3, 6, 9, and 12 post-transplant. At each visit, a physical exam, medication tracking, assessment of graft survival, and blood and urine collection will occur. At the Week 6 and Month 12 visits, intravascular ultrasound and echocardiograms will occur. At the Week 6, Month 6, and Month 12 visits, endomyocardial biopsies will also occur. No immunosuppressive therapy will be provided by the study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 10 and a body mass of 30 kg (66 lbs) or more
* On waiting list for a heart transplant for whom a donor heart available
* Willing to comply with study protocol
* Willing to use acceptable forms of contraception
* Parent or guardian willing to provide consent, if applicable

Exclusion Criteria:

* Receiving multiple organ transplants
* Previously received organ transplants
* Other comorbidities that, in the opinion of the site investigator, would interfere with the study
* Currently taking immunosuppression for nontransplant reasons
* Participation in an interventional clinical trial
* Pregnancy or breastfeeding

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who are on the waiting list for a heart transplant at one of the participating study sites (listed below)
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2007-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Composite Measure of Transplant Health | 12 months after enrollment in study
  A composite of incidence of the following:
  * Death,
  * Re-transplantation or re-listed for transplantation,
  * Biopsy proven acute rejection (BPAR) of > 2R,
  * Episode of rejection associated with hemodynamic compromise,
  * Coronary artery vasculopathy defined by a change in MIT of >0.5 mm between study entry and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S. Heeger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Mohamed H. Sayegh, MD, Principal Investigator — Brigham and Women's Hospital; Randall Starling, MD, Study Chair — The Cleveland Clinic
Locations (12):
- United States (12):
  - University of California, San Francisco, California
  - Northwestern University Medical School, Chicago, Illinois
  - Loyola University School of Medicine, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Utah, LDS Hospital, Salt Lake City, Utah
  - University of Utah, VACM.LDS, Salt Lake City, Utah

REFERENCES:
- [Background] Jiang S, Lechler RI. CD4+CD25+ regulatory T-cell therapy for allergy, autoimmune disease and transplant rejection. Inflamm Allergy Drug Targets. 2006 Dec;5(4):239-42. doi: 10.2174/187152806779010981. PMID 17168794
- [Background] Starling RC, Pham M, Valantine H, Miller L, Eisen H, Rodriguez ER, Taylor DO, Yamani MH, Kobashigawa J, McCurry K, Marboe C, Mehra MR, Zuckerman A, Deng MC; Working Group on Molecular Testing in Cardiac Transplantation. Molecular testing in the management of cardiac transplant recipients: initial clinical experience. J Heart Lung Transplant. 2006 Dec;25(12):1389-95. doi: 10.1016/j.healun.2006.10.002. No abstract available. PMID 17178330
- [Background] Zheng XX, Sanchez-Fueyo A, Sho M, Domenig C, Sayegh MH, Strom TB. Favorably tipping the balance between cytopathic and regulatory T cells to create transplantation tolerance. Immunity. 2003 Oct;19(4):503-14. doi: 10.1016/s1074-7613(03)00259-0. PMID 14563315
- [Result] Starling RC, Stehlik J, Baran DA, Armstrong B, Stone JR, Ikle D, Morrison Y, Bridges ND, Putheti P, Strom TB, Bhasin M, Guleria I, Chandraker A, Sayegh M, Daly KP, Briscoe DM, Heeger PS; CTOT-05 consortium. Multicenter Analysis of Immune Biomarkers and Heart Transplant Outcomes: Results of the Clinical Trials in Organ Transplantation-05 Study. Am J Transplant. 2016 Jan;16(1):121-36. doi: 10.1111/ajt.13422. Epub 2015 Aug 10. PMID 26260101
- See also: Click here for the Clinical Trials in Organ Transplantation [CTOT] public Web site — http://www.ctotstudies.org
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/